CLINICAL TRIAL: NCT03589677
Title: Brain Involvement in Myotonic Dystrophy Type I: From Functional Neuroimaging to the Impact on Quality of Life
Acronym: BrainDM
Status: Completed | Type: Observational
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, prof. Corrado Angelini, professor, M.D., IRCCS San Camillo, Venezia, Italy
Other Study IDs: IRCCSSanCamillo
Record Dates: First submitted 2018-05-10; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Myotonic Dystrophy Type 1 (DM1)
Keywords: DM1; Brain; MRI
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myotonic dystrophy type 1: Subjects of both sexes with a diagnosis of Steinert's disease (DM1), de novo or with the previous diagnosis that shows significant worsening detectable during the follow-up foreseen by the normal cure procedure with clinical presentation indicating a CNS compromise will be evaluated for:
  * quality of life evaluation
  * exam of neuroimaging
  * study of myomiRNAs before and after rehabilitation

SUMMARY:
This project aims to characterize DM1 patients, by collecting clinical, neuropsychological, neuroimaging, and molecular rehabilitative data, in order to elucidate the etiology of cognitive troubles, with special attention to the impact of those dysfunctions on quality of life.

DETAILED DESCRIPTION:
Myotonic Dystrophy Type 1 (DM1), the most common form of muscular dystrophy in adulthood, is characterized by a multisystemic involvement in skeletal muscle (atrophy and progressive hyposthenia, predominantly in the distal districts, and myotonic phenomenon), and of the cardiac, ocular, endocrine, gastrointestinal and central nervous system (CNS) systems. The disease, of a genetic nature, is transmitted as an autosomal dominant trait and is due to an abnormal expansion of the CTG nucleotide triplet of the gene that encodes a kinase protein (DMPK), located on chromosome 19q13.3. Based on the expansion number of nucleotide triplets, 4 classes of expansion were identified: E1, E2, E3, E4, which are directly related to the severity of the phenotype. The pathogenetic basis of the disease is not yet clear to date; however, it is hypothesized that the mutation results in the expression of abnormal RNA transcripts that induce an alteration of the splicing mechanisms of different gene products. The disease frequently presents a typical profile of CNS disorders, characterized by a chronic and progressive pattern. The clinically identifiable symptomatology consists of cognitive disorders (visual-spatial, attention, executive functions), from alterations in the emotional sphere (depressed mood, anxiety and apathetic temperament) and from obsessive / avoiding / passive-aggressive personality traits. A difficulty in recognizing facial emotional states has also been reported. The overall intellectual performance tends to be at the lower limits of the norm when compared to the population of equal age and education. From the neuroradiological point of view, the presence of cortical atrophy, usually more evident in the frontal and temporal, and of white matter lesions spread on both hemispheres, often asymmetric, was detected. Despite the high number of studies on the subject, the frequency and localization of these abnormalities, as well as their relationship to cognitive involvement, the age of onset, duration of disease and genetic profile have not yet been clarified. In clinical practice, patients frequently present a partial impairment of insight, or the psychological ability to have a clear and complete awareness of their condition of illness, the incidence of which, however, has never been investigated. This disorder, also defined by the name of anosognosia, generates in the patient a partial admission of difficulties, which interferes with its adaptability to treatments and in the relationship with the caregiving figures. Lack of awareness about one's state of illness is a psychological condition found in various neurological diseases of an organic or neurodegenerative nature. The neuroanatomical and neuropsychological bases are complex and to date not fully known. The frontal lobes have been identified as possible neuroanatomical localizations of the disorder; however, data in the literature about the relationship between executive function deficits and anosognosia are extremely conflicting. In this patients, the rehabilitative intervention is useful for optimizing muscle tropism and prevents further atrophy of disused muscle fibers. MicroRNAs (miRNAs/miRs) miR-1, miR-206, miR-133a, and miR-133b are called "myomiRs" and are involved in myogenesis, muscle maintenance, and recovery and can be used as possible biomarkers to follow the effectiveness of rehabilitation treatment. There are currently no similar studies on patients with DM1.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years;
* Presence of cognitive disorders declared by the patient or family members spontaneously or at the specific request of the physician, not to compromise the ability to understand and adhere to what is required by the study protocol;
* Suspected leukoencephalopathy;
* Signing of written informed consent.

Exclusion Criteria:

* clinical picture mainly referring to other neurological diseases (eg dementia, stroke outcomes, etc ...)
* incompatibility with the eligibility criteria: subjects with DM1 who do not show symptoms of involvement of the central nervous system; subjects with previous diagnosis.
* impossibility to perform magnetic resonance examinations as they are dangerous for the patient's health;
* patients with severe psychiatric disorders: Axis 1 or 2 of Diagnostic and Statistical Manual of Mental Disorders (DSM IV);
* patients with severe or severe mental retardation: Intelligence Quotient (IQ) at the Wechsler Adult Intelligence Scale (WAIS) <of 45.
* Abuse of alcohol or other psychoactive substances.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: DM1 subjects of both sexes: de novo or with previous diagnosis that show significant worsening detectable during the follow-up foreseen by the normal cure procedure with clinical presentation indicating a CNS compromise. DM1 is frequently characterized by a significant involvement of the CNS, causing cognitive disorders, mood and behavior, varying from case to case.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-07-03 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2015-06-04 (Actual)

PRIMARY OUTCOMES:
Study of quality of life with INQoL test in DM1 patients | Study of quality of life in DM1 patients. Estimated duration: about 15 months
  The Individualized Neuromuscular Quality of Life Questionnaire (INQoL) patients and caregivers' score will be used for define the possible impact of the pathology on the patient's quality of life. Will be used the INQoL Italian version validated in 2010 (Sansone et al. 2010)

SECONDARY OUTCOMES:
Brain MRI neuroimaging in DM1 patients | Estimated duration: about 16 months.
  Brain DM1 neuroimaging examination with MRI T1 sequences will be collected using 1.5 Tesla scanner and analyzed to verified the possible presence of structural brain alteration. T1 sequences will be used to evaluate cortical atrophy in DM1 patients.
Study of circulating myomiRNAs in DM1 patients before and after rehabilitation | Estimated duration: about 16 months.
  New circulating molecular biomarkers, muscle specific-microRNAs (myomiRNAs), will be studied, before and after a period of 6 weeks of rehabilitation protocol, in blood of DM1 patients. MyomiRNAs could be used to evaluate the effect of physical rehabilitation since they appear to be linked to muscle atrophy. Rehabilitation protocol and methodologies have been published and validated by Cudia (Cudia et al.; 2016)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonini G, Mainero C, Romano A, Giubilei F, Ceschin V, Gragnani F, Morino S, Fiorelli M, Soscia F, Di Pasquale A, Caramia F. Cerebral atrophy in myotonic dystrophy: a voxel based morphometric study. J Neurol Neurosurg Psychiatry. 2004 Nov;75(11):1611-3. doi: 10.1136/jnnp.2003.032417. PMID 15489397
- [Background] Antonini G, Soscia F, Giubilei F, De Carolis A, Gragnani F, Morino S, Ruberto A, Tatarelli R. Health-related quality of life in myotonic dystrophy type 1 and its relationship with cognitive and emotional functioning. J Rehabil Med. 2006 May;38(3):181-5. doi: 10.1080/16501970500477967. PMID 16702085
- [Background] Carlesimo GA, Caltagirone C, Gainotti G. The Mental Deterioration Battery: normative data, diagnostic reliability and qualitative analyses of cognitive impairment. The Group for the Standardization of the Mental Deterioration Battery. Eur Neurol. 1996;36(6):378-84. doi: 10.1159/000117297. PMID 8954307
- [Background] Di Costanzo A, Santoro L, de Cristofaro M, Manganelli F, Di Salle F, Tedeschi G. Familial aggregation of white matter lesions in myotonic dystrophy type 1. Neuromuscul Disord. 2008 Apr;18(4):299-305. doi: 10.1016/j.nmd.2008.01.008. Epub 2008 Mar 11. PMID 18337099
- [Background] Meola G, Sansone V. Cerebral involvement in myotonic dystrophies. Muscle Nerve. 2007 Sep;36(3):294-306. doi: 10.1002/mus.20800. PMID 17486579
- [Background] Minnerop M, Weber B, Schoene-Bake JC, Roeske S, Mirbach S, Anspach C, Schneider-Gold C, Betz RC, Helmstaedter C, Tittgemeyer M, Klockgether T, Kornblum C. The brain in myotonic dystrophy 1 and 2: evidence for a predominant white matter disease. Brain. 2011 Dec;134(Pt 12):3530-46. doi: 10.1093/brain/awr299. Epub 2011 Nov 29. PMID 22131273
- [Background] Modoni A, Silvestri G, Vita MG, Quaranta D, Tonali PA, Marra C. Cognitive impairment in myotonic dystrophy type 1 (DM1): a longitudinal follow-up study. J Neurol. 2008 Nov;255(11):1737-42. doi: 10.1007/s00415-008-0017-5. Epub 2008 Sep 24. PMID 18821050
- [Background] Perini GI, Menegazzo E, Ermani M, Zara M, Gemma A, Ferruzza E, Gennarelli M, Angelini C. Cognitive impairment and (CTG)n expansion in myotonic dystrophy patients. Biol Psychiatry. 1999 Aug 1;46(3):425-31. doi: 10.1016/s0006-3223(99)00016-5. PMID 10435210
- [Background] Ries ML, Schmitz TW, Kawahara TN, Torgerson BM, Trivedi MA, Johnson SC. Task-dependent posterior cingulate activation in mild cognitive impairment. Neuroimage. 2006 Jan 15;29(2):485-92. doi: 10.1016/j.neuroimage.2005.07.030. Epub 2005 Aug 15. PMID 16102979
- [Background] Romeo V, Pegoraro E, Ferrati C, Squarzanti F, Soraru G, Palmieri A, Zucchetta P, Antunovic L, Bonifazi E, Novelli G, Trevisan CP, Ermani M, Manara R, Angelini C. Brain involvement in myotonic dystrophies: neuroimaging and neuropsychological comparative study in DM1 and DM2. J Neurol. 2010 Aug;257(8):1246-55. doi: 10.1007/s00415-010-5498-3. Epub 2010 Mar 11. PMID 20221771
- [Background] Gambardella S, Rinaldi F, Lepore SM, Viola A, Loro E, Angelini C, Vergani L, Novelli G, Botta A. Overexpression of microRNA-206 in the skeletal muscle from myotonic dystrophy type 1 patients. J Transl Med. 2010 May 20;8:48. doi: 10.1186/1479-5876-8-48. PMID 20487562
- [Background] Salehi LB, Bonifazi E, Stasio ED, Gennarelli M, Botta A, Vallo L, Iraci R, Massa R, Antonini G, Angelini C, Novelli G. Risk prediction for clinical phenotype in myotonic dystrophy type 1: data from 2,650 patients. Genet Test. 2007 Spring;11(1):84-90. doi: 10.1089/gte.2006.0511. PMID 17394397
- [Background] Salvatori S, Fanin M, Trevisan CP, Furlan S, Reddy S, Nagy JI, Angelini C. Decreased expression of DMPK: correlation with CTG repeat expansion and fibre type composition in myotonic dystrophy type 1. Neurol Sci. 2005 Oct;26(4):235-42. doi: 10.1007/s10072-005-0466-x. PMID 16193250
- [Background] Salvatori S, Furlan S, Fanin M, Picard A, Pastorello E, Romeo V, Trevisan CP, Angelini C. Comparative transcriptional and biochemical studies in muscle of myotonic dystrophies (DM1 and DM2). Neurol Sci. 2009 Jun;30(3):185-92. doi: 10.1007/s10072-009-0048-4. Epub 2009 Mar 27. PMID 19326042
- [Background] Schillings ML, Kalkman JS, Janssen HM, van Engelen BG, Bleijenberg G, Zwarts MJ. Experienced and physiological fatigue in neuromuscular disorders. Clin Neurophysiol. 2007 Feb;118(2):292-300. doi: 10.1016/j.clinph.2006.10.018. Epub 2006 Dec 12. PMID 17166763
- [Background] Sistiaga A, Urreta I, Jodar M, Cobo AM, Emparanza J, Otaegui D, Poza JJ, Merino JJ, Imaz H, Marti-Masso JF, Lopez de Munain A. Cognitive/personality pattern and triplet expansion size in adult myotonic dystrophy type 1 (DM1): CTG repeats, cognition and personality in DM1. Psychol Med. 2010 Mar;40(3):487-95. doi: 10.1017/S0033291709990602. Epub 2009 Jul 23. PMID 19627641
- [Background] Winblad S, Lindberg C, Hansen S. Cognitive deficits and CTG repeat expansion size in classical myotonic dystrophy type 1 (DM1). Behav Brain Funct. 2006 May 15;2:16. doi: 10.1186/1744-9081-2-16. PMID 16696870
- [Background] Winblad S, Hellstrom P, Lindberg C, Hansen S. Facial emotion recognition in myotonic dystrophy type 1 correlates with CTG repeat expansion. J Neurol Neurosurg Psychiatry. 2006 Feb;77(2):219-23. doi: 10.1136/jnnp.2005.070763. PMID 16421126
- [Background] Winblad S, Jensen C, Mansson JE, Samuelsson L, Lindberg C. Depression in Myotonic Dystrophy type 1: clinical and neuronal correlates. Behav Brain Funct. 2010 May 19;6:25. doi: 10.1186/1744-9081-6-25. PMID 20482818
- [Background] Sansone VA, Panzeri M, Montanari M, Apolone G, Gandossini S, Rose MR, Politano L, Solimene C, Siciliano G, Volpi L, Angelini C, Palmieri A, Toscano A, Musumeci O, Mongini T, Vercelli L, Massa R, Panico MB, Grandi M, Meola G. Italian validation of INQoL, a quality of life questionnaire for adults with muscle diseases. Eur J Neurol. 2010 Sep;17(9):1178-1187. doi: 10.1111/j.1468-1331.2010.02992.x. Epub 2010 Mar 30. PMID 20374278
- [Background] Cudia P, Weis L, Baba A, Kiper P, Marcante A, Rossi S, Angelini C, Piccione F. Effects of Functional Electrical Stimulation Lower Extremity Training in Myotonic Dystrophy Type I: A Pilot Controlled Study. Am J Phys Med Rehabil. 2016 Nov;95(11):809-817. doi: 10.1097/PHM.0000000000000497. PMID 27088471